CLINICAL TRIAL: NCT06949735
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Clinical Trial to Investigate the Effect of Digestive Enzyme Supplementation on Postprandial Responses to a High-macronutrient Meal
Brief Title: Clinical Trial on Digestive Enzymes: Effects on Post-Meal Response to High-Macronutrient Meals
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pancap Pharma Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: P02-24-01-T0074
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Digestion; Healthy; Gastrointestinal Wellbeing; Gastrointestinal Supplements
Keywords: Digestive enzyme; Gastrointestinal; Digestion; High-macronutrient meal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digestive Enzyme Blend (Active Comparator): Active ingredients: Porcine Pancreatic Enzyme
  Interventions: Dietary Supplement: Digestive Enzyme Blend
- Placebo (Placebo Comparator): Active ingredients: None
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Digestive Enzyme Blend — Oral
  Arms: Digestive Enzyme Blend
Dietary Supplement: Placebo — Oral
  Arms: Placebo

SUMMARY:
This study aims to show how digestive enzyme supplements help the body break down fats, proteins, and carbohydrates, especially after eating a high-macronutrient meal. Digestive enzymes are essential for nutrient absorption, but some people-such as those with certain medical conditions or high-protein diets-may not produce enough on their own. Poor digestion can lead to bloating, discomfort, and gut imbalances. This clinical trial tests a delayed-release, porcine-derived enzyme blend to see if it improves digestion and reduces symptoms like bloating and gas after eating a high-macronutrient meal.

DETAILED DESCRIPTION:
This study explores the potential benefits of digestive enzyme supplementation for individuals consuming high-macronutrient meals. Digestive enzymes play an important role in breaking down macronutrients to facilitate nutrient absorption. While the body naturally produces these enzymes, certain factors such as genetic predisposition, aging, or high dietary intake of fats and proteins can strain the digestive system, leading to incomplete digestion and gastrointestinal discomfort.

High-macronutrient meals require significant enzymatic activity for proper breakdown, and inadequate digestion can result in symptoms like bloating, indigestion, and changes in gut microbiota. Undigested fats and proteins in the colon can contribute to digestive discomfort, while improperly broken-down carbohydrates may lead to increased gas production and microbial imbalances. These effects can impact overall digestive efficiency, nutrient availability, and gut health.

This clinical trial investigates the efficacy of a delayed-release, porcine-derived enzyme blend containing 20,000 lipase units in improving digestion and gastrointestinal well-being. The study follows a randomized, placebo-controlled, crossover design to assess how this enzyme supplement affects macronutrient breakdown and post-meal symptoms. Researchers will evaluate both immediate effects after a single dose and longer-term benefits after seven days of supplementation, including its impact on quality of life. The findings may provide insight into whether digestive enzyme supplementation can enhance nutrient absorption and alleviate digestive discomfort in individuals consuming high-macronutrient diets.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults who are 18 to 60 years of age (inclusive).

In good general health (no underlying diseases or conditions) as deemed by the investigator.

Have a body mass index (BMI) between 18.5 to 29.9 kg/m2 (inclusive).

Weigh no less than 60 kilograms at screening and baseline.

Self-reported presence of GI symptoms after consuming a high-fat meal.

Are able to orally consume a porcine-based product in a form of capsule.

Are able to consume a high-macronutrient meal within 20 minutes in-clinic, consisting of the following items:

* 1 x BOOST® Protein+ Chocolate Meal Replacement Shake (325 mL)
* 1 x McDonald's Sausage N'Egg McMuffin®
* 1 x 3.25% Whole Milk (~250 mL)
* 2 x McDonald's Hash Brown
* 1 x McDonald's Hotcakes with Butter (no syrup)

Are able to consume a high-macronutrient meal at home each day as per the requirements:

* Supplement participants' meals to ensure the macronutrient targets are met with a supply of CLIF Builders Chocolate Peanut Butter Flavour Protein Bars (~1 per day) prior to the at-home period.
* Consume the high-macronutrient at-home meal within the hours of 11:00 am to 7:00 pm daily.
* At-home meals must be purchased from commonly available fast food restaurants (e.g., McDonald's, Harvey's, Burger King) that provide publicly accessible nutrition information.

Non-smokers (including nicotine vaping) and have not used any nicotine products (patches, gums, etc.) for > 3 months prior to Visit 2.

Non-smoker is defined as someone who does not habitually/regularly use products containing nicotine.

Have a glycated hemoglobin (HbA1c) below 5.7% as assessed at screening.

Agree not to donate blood during the study and within 90 days after completing the study.

Have suitable veins for repeated venipuncture.

Have maintained consistent dietary habits, including medication and supplement intake, and lifestyle for the last 3 months before screening and agree to maintain them throughout the study (with the exception of the high-macronutrient meals).

Agree to follow the restrictions on concomitant treatments

Agree to follow the restrictions on lifestyle

Agree to use acceptable contraceptive methods

Willing and able to agree to the requirements of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

Individuals who are lactating, pregnant or planning to become pregnant during the study, or demonstrate a positive pregnancy test at Visit 2.

Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients, or any of the ingredients in the high-macronutrient meal (in-clinic and at home).

Currently following, or plan to follow a restrictive diet during the study, including low-fat, ketogenic or any other diet that significantly alters macronutrient intake.

Have Type I diabetes, Type II diabetes, high blood pressure (≥140 systolic or ≥90 diastolic mmHg), or thyroid disease.

Have a diagnosis of hypercholesterolemia or hypertriglyceridemia.

Have a history of liver or gallbladder disease or stomach ulcers.

Have a history of irritable bowel syndrome (IBS), inflammatory bowel disease (IBD, including ulcerative colitis), functional constipation or diarrhea (defined by the Rome IV diagnostic criteria), functional dyspepsia, celiac disease, malabsorption, gastroparesis, diverticulosis, gastric or duodenal ulcers, or eating disorder; or have a history of intestinal surgery (excluding appendectomy or herniorrhaphy) or bariatric surgery.

Have blood or bleeding disorders (e.g. anemia).

Have medical condition(s) known to interfere with absorption, distribution, metabolism, or excretion of the study product (e.g., Crohn's disease, short bowel, acute or chronic pancreatitis, or pancreatic insufficiency).

Have a history of heart/cardiovascular disease, renal disease (dialysis or renal failure), hepatic impairment/disease, immune disorders and/or immunocompromised (i.e., HIV/AIDS).

Have a history of cancer (except localized skin cancer without metastases or in situ cervical cancer), unless recovery occurred more than 5 years before the screening visit.

Are receiving treatments for or have been hospitalized in the last 12 months for psychiatric disorders (e.g., depression, bipolar disorder, schizophrenia, etc.).

Reports a clinically significant illness during the 28 days before the first dose of study product.

Major surgery in 3 months prior to screening or planned major surgery during the study.

Have a history of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program) or use that in the opinion of the investigator may be of a concern for the study.

Significant blood loss or blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to first dose of study product or a blood donation of more than 450 mL within 90 days prior to first dose of study product.

Donation of plasma (e.g., plasmapheresis) within 15 days prior to first dose of study product.

Current enrollment or past participation in another study with any product(s) with at least one active ingredient within 28 days before first dose of study product or longer, if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.

Living in the same household as another currently/previously enrolled participant in the present study.

Any other medical condition/situation or use of medications/supplements/therapies that, in the opinion of the investigator, may adversely affect the participant's ability to participate in the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
To Assess the effect of the TP on lipid digestion after a single dose using area under the curve (AUC0-t) - Total Triglycerides | 30,60,90,120,180,210,240,270,300,330 and 360 minutes
  Comparison of total Triglycerides (TG) up to 360 min in response to the high-macronutrient meal.

SECONDARY OUTCOMES:
To assess the effect of the TP on lipid digestion after a single dose using maximum concentration (Cmax): Total Triglycerides | 30,60,90,120,180,210,240,270,300,330 and 360 minutes
  Comparison of total triglycerides up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on lipid digestion after a single dose using time to reach maximum concentration (Tmax) - Total Triglycerides | 30,60,90,120,180,210,240,270,300,330 and 360 minutes
  Comparison of total triglycerides up to 360 min in response to the High-macronutrient meal.
To assess the effect of the TP on protein digestion after a single dose using area under the curve (AUC0-t):Total Free Amino Acids (TFAA) | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of total leucine up to 360 min in response to the High-macronutrient meal.
To assess the effect of the TP on protein digestion after a single dose using maximum concentration (Cmax):Total Free Amino Acids(TFAA) | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of total free amino acids up to 360 min in response to the High-macronutrient meal.
To assess the effect of the TP on protein digestion after a single dose using time to reach maximum concentration (Tmax):Total Free Amino Acids(TFAA) | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of total free amino acids up to 360 min in response to the High-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using area under the curve (AUC0-t): Glucose | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of glucose up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using maximum concentration (Cmax): Glucose | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of glucose up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using time to reach maximum concentration (Tmax): Glucose | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of glucose up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using area under the curve (AUC0-t): Insulin | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of insulin up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using maximum concentration (Cmax): Insulin | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of insulin up to 360 min in response to the high-macronutrient meal.
To assess the effect of the TP on carbohydrate digestion after a single dose using time to reach maximum concentration (Tmax): Insulin | 30,45,60,75,90,105,120,150,180,210,240,270,300,330,360 minutes
  Comparison of insulin up to 360 min in response to the high-macronutrient meal.
To assess the effect of TP on appetite after a single dose using VAS score - Pre dose and Pre Meal | 30,90,120,180,240,300 and 360 minutes
  Change from pre-dose 30,90,120,180,240 and 360 min after the start of high-macronutrient meal.
To assess the effect of TP on gastrointestinal (GI) symptoms after a single dose using VAS score - Pre -Dose and Pre Meal | 30,90,120,180, and 360 minutes
  Change from pre-dose 30,90,120,180, and 360 min after the start of high-macronutrient meal.
To assess the effect of TP on abdominal distention after a single dose in waist Circumference - Pre -Dose and Pre Meal | 30,90,120,180, and 360 minutes
  Change from pre-dose 30,90,120,180, and 360 min after the start of high-macronutrient meal.
To assess the effect of the TP on GI-related quality of life after 7 days of supplementation assessed by the PROMIS Scale V1.1 GI Gas and Bloating | 7 days
  Change from baseline to 7 days in severity rating of GI symptoms.

OTHER OUTCOMES:
To assess the safety of the TP | 8 weeks
  Report of Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Matoski, Study Director — Pancap Pharma Inc.; John Mikhail, Study Chair — Pancap Pharma Inc.
Locations (1):
- Apex Trials, Guelph, Ontario - on, Canada

IPD SHARING:
Plan to Share IPD: No